CLINICAL TRIAL: NCT00960635
Title: Immunointervention With 1,25-dihydroxy-vitamin D3 in New-onset Type 1 Diabetes
Brief Title: Immunointervention With Calcitriol in New-Onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fur Diabetesforschung, Munich, Germany (Other)
Responsible Party: Anette Ziegler, MD, Institut fuer Diabetesforschung
Purpose: Prevention
Other Study IDs: 336/00
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Type 1 Diabetes
Keywords: new-onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- calcitriol (Active Comparator)
  Interventions: Drug: 1,25-dihydroxy-vitamin D3 (calcitriol)
- pill without agent (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 1,25-dihydroxy-vitamin D3 (calcitriol)
  Arms: calcitriol
Drug: placebo — pill without agent
  Arms: pill without agent

SUMMARY:
This is a randomized, two-arm, placebo-controlled phase-2 trial to determine whether the daily intake of 1,25-dihydroxy-vitamin D3 [1,25(OH)2D3], improves beta cell function in patients with recently diagnosed type 1 diabetes. The treatment consists of the daily oral administration of 0.25 µg 1,25(OH)2D3 or placebo for 9 months and an equal follow-up time without supplementation. Fasting, peak and AUC C-peptide concentrations during a 2-hour mixed meal tolerance test are measured at the beginning of the study, as well as at the end of the treatment and the follow-up period in month 9 and 18. The null hypothesis is that there is no difference between 1,25(OH)2D3 treated subjects and the placebo group in the AUC C-peptide at month 18.

ELIGIBILITY:
Inclusion Criteria:

* New onset Typ 1 diabetes (< 6 weeks insulin therapy)
* Age 18-39 years
* GADA and/or IA-2A positive

Exclusion Criteria:

* Kidney disease
* Pregnancy
* Lactating

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Dates: Start 2001-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anette G Ziegler, MD, Principal Investigator — Institut fuer Diabetesforschung
Locations (1):
- Institut fuer Diabetesforschung, Munich, Germany

REFERENCES:
- [Derived] Walter M, Kaupper T, Adler K, Foersch J, Bonifacio E, Ziegler AG. No effect of the 1alpha,25-dihydroxyvitamin D3 on beta-cell residual function and insulin requirement in adults with new-onset type 1 diabetes. Diabetes Care. 2010 Jul;33(7):1443-8. doi: 10.2337/dc09-2297. Epub 2010 Mar 31. PMID 20357369